CLINICAL TRIAL: NCT03363672
Title: Evaluation of the Prevalence and Impact of Chronic Postoperative Pain and Risk Factor Analysis: a Multi-center Prospective Cohort Study
Brief Title: Prevalence, Impact and Predictors of Chronic Postoperative Pain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Huang YuGuang, Chairman of anesthesisology department, Peking Union Medical College Hospital
Other Study IDs: PUMCH-CPP
Record Dates: First submitted 2017-11-20; First posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: Chronic Postoperative Pain
Keywords: Chronic Postoperative Pain; Daily Life; Risk Factor
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 48 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients receiving surgery: No intervention will be administered. Patients included will be asked to return a questionnaire regarding chronic postoperative pain via app.

SUMMARY:
Chronic postoperative pain (CPP) remains a disturbing and obscure clinical problem, which could last for more than 3 months after surgery. The aim of present study was to assess the prevalence of CPP, investigate its impact on life quality and explore its potential risk factors. After informed consent was signed, patients receiving surgery under general anesthesia in Peking Union Medical College Hospital and other medical centers participating in this study during 2018 will be included. Patients' preoperative information will be collected from medical record, including basic demographic data, primary disease and previous chronic diseases. Intraoperative information will be obtained from anesthesia record, including surgical scope, duration, length and location of incisions and blood loss. Acute pain will be evaluated in the ward of the department of surgery, when an app will be installed on patients' mobile phones. Our long-term postoperative follow-up would be performed by sending out survey questionnaires via this app in the 4th, 8th, 16th, 32th, and 48th weeks after surgery. The survey covers questions regarding the intensity, characteristic, location and impact on daily activities of CPP. Information regarding treatment of CPP will also be collected, if any. All the data gained will be summarized in our database and analyzed.

DETAILED DESCRIPTION:
Chronic postoperative pain (CPP) remains a disturbing and obscure clinical problem, which could persist beyond wound healing phase and last for more than 3 months after surgery. The prevalence of CPP after sternotomy is estimated to be as high as 14%-61%, according to several recent studies. However, CPP following other types of surgeries has not been well evaluated. There is paucity of literature regarding the impact of CPP on daily life as well. Additionally, the identification of predisposing factors for CPP would provide clues for its prevention and treatment. The aim of present study was to assess the prevalence of CPP, investigate its impact on life quality and explore its potential risk factors.

After informed consent was signed, patients receiving surgery under general anesthesia during 2018 will be included. The sample size in Peking Union Medical College Hospital is estimated to be approximately 700. Furthermore, we are trying to contact with other large hospitals in China to make a multi-center study.

Patients' preoperative information will be collected from medical record, including basic demographic data, primary disease (tumor size, location and peripheral invasion) and previous chronic diseases (hypertension, diabetes, coronary heart disease, chronic kidney disease, anxiety and depression). Intraoperative information will be obtained from anesthesia record, including surgical scope, duration, length and location of incisions and blood loss. Postoperative pain control methods can be learned from medical orders. Acute pain will be evaluated in the ward of the department of surgery before discharge. At the same time, an app will be installed on patients' mobile phones. Our long-term postoperative follow-up would be performed by sending out survey questionnaires via this app in the 4th, 8th, 16th, 32th, and 48th weeks after surgery. The survey covers questions regarding the intensity (Wong-Baker FACES Pain Rating Scale), characteristic, location and impact on daily activities (Brief Pain Index, BPI) of CPP. Furthermore, information regarding treatment of CPP will also be collected, if any. All the data obtained from app could be included into our database and statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving surgery under general anesthesia during 2018 in Peking Union Medical College Hospital and other medical centers participating in this study.
* Aged 18-70 years.

Exclusion Criteria:

* Previous surgery history;
* Preoperative chronic pain history;
* Injury;
* Have no access to mobile phone or website;
* Postoperative chronic infection;
* Non-radical incision of tumor or malignancy recurrence during follow-up;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving surgery under general anesthesia during 2018 in Peking Union Medical College Hospital and other medical centers participating in this study
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
The prevalence of chronic postoperative pain | 24 weeks postoperatively
  The prevalence of chronic postoperative pain reported by the included patients in the questionnaire issued by app

SECONDARY OUTCOMES:
The prevalence of chronic postoperative pain | 4,8,12,16,20,32,40,48 weeks postoperatively
  The prevalence of chronic postoperative pain reported by the included patients in the questionnaire issued by app
Wong-Baker Faces Pain Rating Scale | 4,8,12,16,20,24,32,40,48 weeks postoperatively
  The intensity of CPP will be evaluated by Wong-Baker FACES Pain Rating. The scale shows a series of faces ranging from a happy face at 0 which represents "no hurt" to a crying face at 10 which represents "hurts worst." Scale.
Characteristics and location of chronic postoperative pain | 4,8,12,16,20,24,32,40,48 weeks postoperatively
  The common characteristics and location of CPP will also be summarized according to the patients' choice in survey.
Brief Pain Index | 4,8,12,16,20,24,32,40,48 weeks postoperatively
  Brief Pain Index will be used to assess the impact of chronic postoperative pain on daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Yuguang Huang, MD., Study Chair — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared via a database.
Time Frame: IPD will become available from 2018-1-1 to 2019-12-31.
Access Criteria: All the IPD will be included in a public database shared by all the medical centers participating in this study.